CLINICAL TRIAL: NCT07307209
Title: A Comparative Evaluation of Whole Maxillary Dentition Distalization Using Sliding Jig vs. Retraction Hooks Anchored by IZC Miniscrews: A Randomized Clinical Trial
Brief Title: "Sliding Jigs vs Retraction Hooks for Maxillary Dentition Distalization Using IZC Miniscrews"
Acronym: SJRH-IZC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Dr. Nagi Alawdi, Researcher, Sana'a University, Sana'a University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-ORTHO-IZC-RCT-2025; EC-OR: 03\9\ 2025 (Other: Sana'a University medical Ethics Committee)
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Skeletal Class II Malocclusion
Keywords: Maxillary Distalization; IZC Miniscrew; Sliding Jig

STUDY DESIGN:
Intervention Model Description: This is a randomized interventional clinical trial comparing two orthodontic mechanics for whole maxillary dentition distalization using infrazygomatic crest miniscrews in Class II patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sliding Jig (Experimental): Description: Participants in this group will undergo whole maxillary dentition distalization using Sliding Jig mechanics anchored by infrazygomatic crest (IZC) miniscrews.
  Interventions: Device: Sliding jig
- Retraction Hook (Active Comparator): Description: Participants in this group will undergo whole maxillary dentition distalization using Retraction Hooks mechanics anchored by infrazygomatic crest (IZC) miniscrews.
  Interventions: Device: retraction hooks

INTERVENTIONS:
Device: Sliding jig — participants in this group will undergo whole maxillary dentition distalization using Sliding Jig mechanics anchored by infrazygomatic crest (IZC) miniscrews.
  Arms: Sliding Jig
Device: retraction hooks — participants in this group will undergo whole maxillary dentition distalization using Retraction Hooks mechanics anchored by infrazygomatic crest (IZC) miniscrews.
  Arms: Retraction Hook

SUMMARY:
This randomized controlled clinical trial aims to compare the clinical efficacy, efficiency, and biomechanical differences between two methods for total maxillary dentition distalization: (1) the use of a Sliding Jig and (2) the use of Retraction Hooks, both anchored by Infrazygomatic Crest (IZC) miniscrews. The study will assess rates of distalization, anchorage loss, dentoalveolar tipping, patient comfort, and treatment-associated side effects.

DETAILED DESCRIPTION:
Background and Rationale In non-extraction orthodontic treatment of Class II malocclusion or maxillary dentoalveolar protrusion, whole maxillary dentition distalization is a key treatment modality. The advent of temporary anchorage devices (TADs), specifically infrazygomatic crest (IZC) miniscrews, has revolutionized this approach by enabling predictable posterior translation of the entire maxillary arch without significant anchorage loss or reliance on patient compliance.

However, the biomechanical method for transferring force from the miniscrew to the dentition-whether through a sliding jig (continuous force via a rigid attachment) or separate retraction hooks (segmented force applied to individual teeth or groups)-may lead to clinically significant differences in movement type, efficiency, stability, and patient experience. No randomized clinical trial to date has directly compared these two popular clinical approaches.

This study will provide evidence-based recommendations for optimizing clinical mechanics in whole arch distalization protocols.

Objectives Primary Objective To compare the rate of maxillary first molar distalization (in mm/month) achieved using the sliding jig technique versus retraction hooks anchored by IZC miniscrews.

Secondary Objectives To assess the amount and type of tooth movement (tipping vs. translation) of the maxillary first molars and central incisors.

To evaluate anchorage stability by measuring 3D positional changes of the IZC miniscrews and any unintended distal movement of the maxillary dentition.

To compare changes in occlusal plane inclination and vertical dentoalveolar effects.

To record and compare patient-reported outcomes, including pain/discomfort levels, oral hygiene difficulty, and appliance interference.

To document clinical side effects, such as miniscrew stability, soft tissue irritation, and root proximity.

Study Design Design: Prospective, parallel-group, randomized controlled clinical trial (RCT).

Allocation Ratio: 1:1. Blinding: Single-blind (Outcome assessor will be blinded to group assignment. Patients and treating clinicians cannot be blinded due to the nature of the intervention). Methodology Participant Selection Source: Patients seeking orthodontic treatment at [Sana'a university]. Sample Size: [To be calculated based on power analysis; e.g., n=20 per group, total N=40].

Randomization & Intervention After consent and initial records, participants will be randomly assigned to Group A (Sliding Jig) or Group B (Retraction Hooks) using computer-generated random numbers in sealed opaque envelopes.

Preintervention records were taken as T0, which include intraoral and extraoral photographs, lateral cephalometric and panoramic radiographs, and study models.

The IZCMI (infra-zygomatic mini-implant) will be 2 × 12 mm in diameter and length, respectively, will be placed in infrazygomatic crest area bilaterally.

The IZCMI will be placed distal to the maxillary first molar at 11-12 mm above the cemento-enamel junction at an angle of 50-70° from the occlusal plane.

Retraction hooks were modeled using 0.036-inch crimpable hook stainless steel (soldered 23-gauge stainless steel wire (0.574 mm) for making the hook) and located bilaterally between the lateral incisors and canines. Crimpable hook height of 8 mm will place on the arch wire between the lateral incisors and canines after levelling aligning in one side, and on the other side, A 0.7-mm round SS wire was used to construct the distalization jig. Regarding the design, the distal extension of the jig will be fitted before the molar band or tube. The mesial extension had a helix that surrounded the main archwire, and the jig in the distal section had a lever arm distal to the canine. The lever arm will be set at height according to the mini screw and center of resistance height.

For en-masse anterior retraction, according to Wu et al. a force of 300 g will be given from the IZC screws to the crimpable hooks placed in the region between lateral incisors and canines, and to the lever arm of sliding jig distal to the canine through nickel-titanium (NiTi) closed coil springs/E chains, which activated every 4 weeks. The amount of force was measured using a dontrix gauge.

All patients will be treated using a pre-adjusted edgewise appliance system using a Roth prescription, a slot size of 0.022 × 0.028 inch, and metal brackets with conventional ligation. After leveling and aligning the dentition, stainless steel wire (0.019 x 0.025 inch) was used as the working archwire for the maxillary dentition distalization and ended when an acceptable overjet will be achieved, and on reaching Class I relationship molar and canine.

For all patient, miniscrews will be checked for stability, every 4 weeks intra-oral scanning will be taken. Use digital scans to create 3D models of the dental arch and measure maxillary dentation movement with precision. The 3D model images will be assessed using Orth Analyzer software (3Shape, Copenhagen, Denmark). Furthermore, scanned 3D models will be superimposed over the subsequent model to measure the average monthly distalization. Anchorage loss of the first maxillary molars will be also measured on the digitally scanned models. Furthermore, molar rotation will be measured.

Outcome Measures & Data Collection Primary Outcome: Rate of Molar Distalization. Measured on digital models (from intraoral scans) by comparing the 3D position of the maxillary first molar (mesial contact point) relative to the stable palatal rugae at T0 (pre-distalization) and T1 (after 4mm distalization achieved or 6 months).

Secondary Outcomes:

Tooth Movement Type: Angular changes (tipping) of molars and incisors on lateral cephalograms.

Anchorage Loss: 3D movement of miniscrews and mandibular molar position (digital models analysis).

Occlusal Plane Change: Cephalometric analysis. Patient-Reported Outcomes: Visual Analog Scale (VAS) for pain/discomfort at 24h, 3d, 7d; questionnaire on oral hygiene and function.

Clinical Side Effects: Miniscrew mobility, inflammation, mucosal coverage (clinical exam).

Reliability Analysis To determine inter-examiner reliability, two examiners will evaluate the images independently. Calibration of the examiners will be undertaken until intra-examiner reliability and reproducibility will be achieved. Kappa statistics will be used for assessing the agreement between observers using the statistical software.

Statistical Analysis:

Data will be evaluated using statistical package SPSS software system, (SPSS Inc, Chicago, Illinois, United States), and descriptive statistical analysis (mean, standard deviation) will be used to obtain the mean and standard deviation for continuous data. Paired t-test will be performed to analyze the changes in pre- and post-distalization. For any of the used tests, results will be considered as statistically significant if p value≤ 0.050.

. Ethical Approval:

* The study protocol will be submitted to the Ethical Committee of the College of Dentistry University of Sana'a, for review and approval.
* Written informed consent will be obtained from the patients of all participants prior to enrollment in the study.
* The study will adhere to the guidelines outlined in the World Medical Association Declaration of Helsinki, ensuring that the research complies with ethical standards for studies involving human subjects.

Expected Significance and Impact This study will provide high-level evidence (Level 2, RCT) to guide clinical decision-making in biomechanics for total arch distalization. Findings will help clinicians choose the most efficient, predictable, and patient-friendly method, ultimately improving treatment quality and efficiency. The results will be disseminated through peer-reviewed publication and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be the following: Adult patients with class II malocclusion (>14 years), present of all permanent teeth fully erupted, Bilateral Class II molar relationship skeletal malocclusion, moderate maxillary arch crowding (less than 5 mm) with maxillary protrusion, absence of craniofacial syndrome. and, except third molars

Exclusion Criteria:

* The subjects having the following conditions will be excluded from the study (1) Patients with transverse dental or skeletal discrepancies. (2) Patients indicated for extraction treatment (except for third molars) or unilateral distalisation treatment (3) Patients with Vertical growth pattern, (4) Patients having periodontal disease, (5) Patients with previous orthodontic treatment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Molar Distalization. | From baseline (start of distalization) to the completion of distalization (an average of 5 months).
  Measured on digital models (from intraoral scans) by comparing the 3D position of the maxillary first molar (mesial contact point) relative to the stable palatal rugae at T0 (pre-distalization) and T1 (after 4mm distalization achieved or 6 months).
Rate of maxillary first molar distalization | From baseline (start of active distalization forces) to the completion of planned distalization (target: 4-6 mm) or at 6 months, whichever comes first.*
  The linear distal movement of the maxillary first molar, measured via 3D superimposition of serial digital intraoral scans on the stable palatal rugae, divided by the active treatment time in months to yield a rate in mm/month.

CONTACTS AND LOCATIONS:
Overall Officials: Nagi H Alawdi, MSc., Principal Investigator — Faculty of Dentistry, Sana'a University; Fuad Luft Almutareb, prf., Study Director — Faculty of Dentistry, Sana'a University
Locations (1):
- Orthodontic department-faculty of dentistry- Sana'a univeristy, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified participant data will be made available:
  Cephalometric measurements, 3D casts, treatment outcomes. For researchers with approved proposals,Within 6 months after publication of results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Supporting information to be shared includes: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), and Analytic Code. Data and supporting documents will become available within 6 months after publication of the study results and will remain accessible for 5 years.
Access Criteria: Individual participant data and supporting documents will be available to researchers who submit a methodologically sound proposal for secondary analyses. Requests will be reviewed and approved by the Principal Investigator. A data sharing agreement must be signed to ensure privacy and ethical use of the data.
URL: https://mailto:nagialawdi@hotmail.com